CLINICAL TRIAL: NCT04100681
Title: Intermittent Negative Pressure to Improve Peripheral Blood Flow in Patients With Peripheral Artery Disease and Intermittent Claudication
Brief Title: Intermittent Negative Pressure; Impact on Peripheral Artery Disease and Intermittent Claudication
Acronym: FlowOx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to slow recruitment and inability to recruit patients during the Covid-19 situation.
Sponsor: Otivio AS (Industry)
Collaborators: mediq Innovation Experts GmbH (Unknown); Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OT-FO-IC
Record Dates: First submitted 2019-09-05; First posted 2019-09-24 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Vascular Disease; Intermittent Claudication; Walking, Difficulty; Critical Limb Ischemia; Ischemia Limb
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication; Mobility Limitation; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: A multi-centre, randomized, sham (placebo) device-controlled, double-blinded trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active FlowOx™ (Active Comparator): The application of pulsating negative pressure will be up to 120 minutes long per day. The pulsating negative pressure used will be approximately 40 mm Hg alternating with ambient air pressure, the pulse consisting of 10 seconds of negative pressure followed by 7 seconds of atmospheric pressure.
  Interventions: Device: Active FlowOx™
- Sham FlowOx™ (Placebo) (Sham Comparator): The application of a mild pulsating negative pressure will be up to 120 minutes long. The pulsating negative pressure used will be approximately 10 mm Hg alternating with ambient air pressure, the pulse consisting of 10 seconds of negative pressure followed by 7 seconds of atmospheric pressure.
  Interventions: Device: Sham FlowOx™ (Placebo)

INTERVENTIONS:
Device: Active FlowOx™ — Treatment is done by the patient at home for about 2 hours per day. Recommended to be 1 hour in the morning and 1 hour in the afternoon.
  Arms: Active FlowOx™
Device: Sham FlowOx™ (Placebo) — Treatment is done by the patient at home for about 2 hours per day. Recommended to be 1 hour in the morning and 1 hour in the afternoon.
  Arms: Sham FlowOx™ (Placebo)

SUMMARY:
The objective is to ensure the pro-active collection of information on quality, safety and performance of FlowOx™ after it is placed on the market. The study will be carried out in a patient population with peripheral artery disease (claudicatio intermittens) to confirm its usefulness and in particular gather information for further improvements of the device related to this patient population. The data collected from the use of the CE-marked FlowOX™ device are change of walking distance, quality of life, and the patient's compliance.

DETAILED DESCRIPTION:
A multi-center, randomized, sham (placebo)-controlled, double-blind trial to assess the efficacy and safety of FlowOx. This is done by comparing the increase in pain free walking distance compared to sham (placebo) device in patients with peripheral arterial disease (PAD) and intermittent claudication.

This study is conducted to assess the efficacy and safety of FlowOx™ compared to a sham FlowOx™ (placebo) device treatment. FlowOx™ can provide intermittent negative pressure (up to - 40 mmHg INP [intermittent negative pressure]) which is known to improve blood flow. The same device will also work as a sham (placebo) device by less negative pressure exerted by the device (in the range of -10 mmHg).

Daily home use of FlowOx™ for 2 hours (divided into minimum two sessions of 1 hour) per day in PAD-patients with intermittent claudication (stage II acc.to EMA, equivalent to Fontaine stage IIb in Germany) relative to sham (placebo) will be provided over a period of 12 weeks.

This efficacy study is evaluating the clinical effects of INP on patient with intermittent claudication with special focus on changes in pain free walking distance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, age greater or equal 18 years
* Stable evidence based pAVK therapy for at least 3 months
* Ability to perform a treadmill test
* Confirmation of clinical diagnosis of PAD as objective evidence of Fontaine stage IIb PAD i.e.:

  * Reduced ankle systolic blood pressure (ABI <0.9) on target leg
  * Pain free walking distance < 200 m in standardized walking test (initial claudication distance (ICD))
* Completion of at least two treadmill tests within a time interval of greater or equal to 1 week prior to randomisation. Maximum change in claudication should not exceed a predefined threshold (<25% for the absolute claudication distance (ACD)).
* Intermittent claudication lasting for at least 3 months
* Stable smoking habits for at least 3 months prior to inclusion
* Signed Informed Consent

Exclusion Criteria:

* PAOD-patients with critical limb ischemia (CLI), equivalent to EMA's or Fontaine's PAOD-stages III and IV
* Any kind of revascularization (endovascular, surgical) in the iliac or other leg arteries within 3 months prior to Visit 1
* Patients with polyneuropathy
* Other illnesses limiting exercise capacity (angina pectoris, heart failure, respiratory disease, orthopedic disease, neurological disorders)
* Use of confounding medications within the last 4 weeks prior the Visit 1 e.g. vasoactive compounds like Cilostazol or Naftidrofuryl
* Uncontrolled hypertension (> 180/95 mmHg) or hypotension (supine < 100 mmHg)
* Severe anemia
* Pregnancy or lactation period
* Woman with childbearing potential without an effective contraceptive method (effective contraception method: hormonal contraceptive, hormonal vaginal devices or injections with prolonged release; an intrauterine device, or a barrier method of contraception such as condom or occlusive cap with spermicide (foam/gel/film/cream/suppository)
* Planned surgical intervention requiring hospitalization during the clinical trial
* Previous inclusion in the present clinical trial or parallel participation in other clinical trials (up to 8 weeks before Visit 1)
* Incapability of understanding nature, meaning and consequences of the clinical trial
* Patient unable to read and or write
* Patients in custody by juridical or official order
* Patients, who are members of the staff of the trial centre, staff of the sponsor or involved Clinical Research Organizations (CRO's), the investigator him-/herself or close relatives of the investigator
* Patients unable to don or doff the FlowOx device (either themselves or with assistance from a helper).
* Diagnosed acute deep vein thrombosis
* Systemic infection
* Alcohol disease or drug abuse
* Malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in pain-free walking distance from baseline to week 12 | baseline to week 12
  The change will be calculated as difference in meters and compared between the interventional and the sham group.

SECONDARY OUTCOMES:
Change in maximal walking distance from baseline to week 12 | 3 months treatment
  The change will be calculated as difference in meters and compared between the interventional and the sham group.
Change in Ankle Brachial index from baseline to week 12 | from baseline to week 12
  Determination of the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium)
Change in Quality of Life from baseline to week 12: EQ-5D-5L | from baseline to week 12
  The 5-level EQ-5D (EuroQol- 5 Dimension) version (EQ-5D-5L) essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  EQ-5D-5L describes the health condition of adults in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). Patient indicate their health states by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ-VAS score is read on a scale of 0-100 points (scale name: health condition), depending on where the patient has set his mark. 0 points mean the worst possible health condition, while 100 points is the best health possible.
Change in activity of daily living from baseline to week 12 | from baseline to week 12
  To evaluate the activity of daily living the standardized questionnaire VascuQoL-6 is used which comprises a set of 6 questions. Each question is scored 1-4. The sum of each individual question score is used to generate a "Total" Score. A higher value indicates better health status.
Determination of compliance of subjects as assessed by the time the device has been running | at week 12
  The FlowOx device records the time the device has been running each time it was started. This record is saved on an USB stick which is readable by the study personnel only and serves to document the patient's compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Lawall, Dr. Med, Principal Investigator — Gemeinschaftspraxis; Silke Zimmermann, Dr. rer.nat., Study Director — HCTC-KKS - Coordinating Center for Clinical Studies
Locations (5):
- Germany (5):
  - Franziskus-Krankenhaus Berlin, Berlin
  - Evangelisches Krankenhaus Hubertus, Gefäßzentrums Berlin-Brandenburg, Berlin
  - Gemeinschaftspraxis, Ettlingen
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Universitätsmedizin Johannes Gutenberg Universität, Mainz

IPD SHARING:
Plan to Share IPD: No